CLINICAL TRIAL: NCT02904785
Title: The Efficacy of Extracorporeal Focused Shock Wave Therapy for Patients With Primary Knee Osteoarthritis
Brief Title: Extracorporeal Focused Shock Wave Therapy for Primary Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Linamara Rizzo Battistella, MD PhD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54013616.1.0000.0068
Record Dates: First submitted 2016-06-29; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Unilateral Primary Osteoarthritis of Knee
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extracorporeal Shock Waves (Experimental): Focused shock waves delivered by an electromagnetic generator with a focus of 5.0cm deep on the affected knee in three different positions. A total of 7000 pulses will be delivered on a weekly session for four weeks.
  Interventions: Device: Extracorporeal Shock Waves; Other: Physical activities
- Sham Extracorporeal Shock Waves (Sham Comparator): Sham focused shock waves delivered by an electromagnetic generator on the affected knee in three different positions. A total of 7000 pulses will be delivered on a weekly session for four weeks. A foam will be placed in the probe as to stop the energy to be transmitted to the patient's knee, so no focused shockwaves will be delivered.
  Interventions: Device: Sham Extracorporeal Shock Waves; Other: Physical activities

INTERVENTIONS:
Device: Extracorporeal Shock Waves
  Arms: Extracorporeal Shock Waves
Device: Sham Extracorporeal Shock Waves
  Arms: Sham Extracorporeal Shock Waves
Other: Physical activities — Patients receive instructions for physical activities for strengthening of femoral quadriceps and stretching of hamstring muscles.

SUMMARY:
The purpose of this study is to determine whether Extracorporeal Focused Shock Wave Therapy reduces knee pain and enhance function in patients with primary knee osteoarthritis.

DETAILED DESCRIPTION:
This study is a placebo controlled Randomized Clinical Trial (RCT) in which the primary outcome is to determine whether Extracorporeal Focused Shock Wave Therapy (ESWT) reduces knee pain comparing the VAS at baseline and one month after the end of the treatment. Function assessment and progression of pain along the treatment are the secondary outcomes. Function will be assessed with the Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC), the Lequesne's Algofunctional Questionnaire for Osteoarthritis of Knee (Lequesne) and the Timed up and Go (TUG).

The ESWT applications will be performed once a week for four consecutive weeks, the patients will be assessed for pain and function before the beginning of the treatment and one week after every application of the ESWT.

The treatment groups will be randomized. The allocation of the patients is sealed and will not be disclosed to the patients nor to the evaluators.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiologic diagnosis of primary knee osteoarthritis (Kellgren & Lawrence I, II or III);
* Capability to understand the Informed Consent Form;
* Chronic pain for at least 3 months prior to inclusion, measured by VAS. (VAS 4 or above);
* Absence of skin injures, infections or tumor in the target knee;
* Availability to comply with the visits.

Exclusion Criteria:

* History of spinal cord stenosis or clinical symptoms of lumbar radiculopathy;
* History or onset neurological diseases;
* Generalized pain or fibromyalgia;
* Inability to walk;
* History of knee surgery in the target knee;
* Secondary causes of osteoarthritis;
* Use of statins and quinolones in the previous year;
* Uncontrolled and ongoing psychiatric diseases;
* Invasive knee treatments with hyaluronic acid infusion, corticosteroids and anaesthetics, in the target knee, up to 6 months previous to study inclusion.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Knee Pain after one month | One month
  Mean change in Visual Analogue Scale (VAS) score one month after the end of the treatment compared to baseline.

SECONDARY OUTCOMES:
Knee pain progression | One week after each of four weekly ESWT applications
  Mean change in VAS score one week after each application compared to baseline.
Knee Pain after three months | Three months
  Mean change in VAS score three months after the end of the treatment compared to baseline.
Lequesne Knee Function progression | One week after each of four weekly ESWT applications
  Mean change in Lequesne score one week after each application compared to baseline.
Lequesne Knee Function after three months | Three months
  Mean change in Lequesne three months after the end of the treatment compared to baseline.
WOMAC Knee Function progression | One week after each of four weekly ESWT applications
  Mean change in WOMAC score one week after each application compared to baseline.
TUG Knee Function progression | One week after each of four weekly ESWT applications
  Mean change in TUG score one week after each application compared to baseline.
WOMAC Knee Function after three months | Three months
  Mean change in WOMAC score three months after the end of the treatment compared to baseline.
TUG Knee Function after three months | Three months
  Mean change in TUG score three months after the end of the treatment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Linamara R Battistella, PhD, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Centro de Pesquisa Clínica do Instituto de Medicina Física e Reabilitação do HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided